CLINICAL TRIAL: NCT03474406
Title: The Effectiveness of Cancer Pain Management Including Early Pain Intervention, Early Multi Modality Treatment and Closed Follow up in Siriraj Outpatient Pain Clinic
Brief Title: The Effectiveness of Cancer Pain Management in Siriraj Outpatient Pain Clinic
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si 622/2017
Record Dates: First submitted 2018-02-18; First posted 2018-03-22 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Pain, Chronic; Cancer
MeSH Terms: conditions — Chronic Pain; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: follow up system and multimodality approach — To provide a new service system for cancer pain in pain clinic by early detecting red flag sign to consult other departments, early alleviating severe pain, following patients intensively by telephone call and giving pain education

SUMMARY:
-Background: Cancer is one of the most common cause of death. Cancer pain is often cited as one of the most feared in cancer patients. Although, WHO guidelines have been provided to improve pain outcome, the results are still unsatisfied. In order to improve cancer pain management we consider to contribute a new guideline which includes interdisciplinary approach, early doing the pain interventions, breakthrough pain, education, high quality of pain assessment and contribute the effectiveness follow-up system

DETAILED DESCRIPTION:
* Objectives:Primary outcome is study the effectiveness of new approach and closed follow up system by relief pain intensity 30% at 3 month up to 80% of all new cancer pain patients in OPD setting Secondary outcomes are quality of life (BPI,ESAS), side effect of treatments and the contributing factors that impact on the outcomes
* Study design:A prospective observational study
* Sample size : 150
* Data collection: General information: age, gender, body weight, height, religion, residence, care giver, occupation, income, education, medical problem Clinical pain information: primary diagnosis, staging, cancer site, current medications Clinical assessment: at three study time points: baseline (initial assessment) and the three subsequent follow-ups (FU1, FU2 and FU3)

ELIGIBILITY:
Inclusion Criteria:

* Cancer pain patients
* more than 18 years old

Exclusion Criteria:

* Clinical instability
* Cannot read and write
* Do not know the diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The new patients with cancer pain in Siriraj outpatients pain clinic
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pain Clinic Siriraj Hospital, Principal Investigator — Mahidol University
Locations (1):
- Faculty of medicine Siriraj Hospital Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited cancer patients who received a new consult for cancer pain at the Siriraj Pain Clinic from January to December 2018. Written informed consent was obtained from all patients
Groups:
- Cancer Patients: Cancer patients 18 years and older who received a new consult for cancer pain at the Siriraj Pain Clinic from January to December 2018. Written informed consent was obtained from all patients. We excluded patients who had difficulties with listening, reading, and writing Thai and those who were unable to interpret the evaluation form/questionnaires.
Period: Overall Study
Arm/Group | Cancer Patients
Started | 150
Completed | 72
Not Completed | 78

BASELINE CHARACTERISTICS:
Arm/Group | Cancer Patients
Number analyzed (Participants) | 150
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [50 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 150
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Thailand | 150
BMI (Body Mass Index) [Median (Inter-Quartile Range); unit: kg/m^2] | 20.7 [18.4 to 23.3]
Marital status [Count of Participants; unit: Participants]
  Married | 105
  Single/Divorce/Widow | 45
Living with [Count of Participants; unit: Participants]
  Family/Sibling | 143
  Alone | 7
Education [Count of Participants; unit: Participants]
  High school and below | 94
  Higher than high school | 56
Numerical Rating Pain scale (0-10: 0 designating no pain, 10 designating worst possible pain) [Median (Inter-Quartile Range); unit: units on a scale] | 5 [4 to 6]
Karnofsky Performance status (KPS) evaluated Functional impairment [Median (Inter-Quartile Range); unit: Percent] — (Karnofsky Performance Status (0-100); 100% indicates no functional impairment, no evident disease, 0% indicates death)
  Percent | 70 [60 to 80]
Cancer status [Count of Participants; unit: Participants]
  Local | 29
  Advanced | 121
Primary tumor [Count of Participants; unit: Participants]
  Gastrointestinal | 40
  Bronchus and lung | 19
  Breast | 9
  Head and neck | 40
  Hematological | 4
  Gynecological | 22
  Urological | 12
  Musculoskeletal | 4
Pain medication taken [Number; unit: participants]
  Opioids | 128
  Acetaminophen | 70
  NSAIDs | 14
  Anticonvulsants | 57
  Antidepressants | 21
  Laxatives | 53
  Antiemetics | 10
Morphine Equivalent Diary Dosage [Median (Inter-Quartile Range); unit: mg/day] | 20 [10 to 31]
History of radiation before study [Count of Participants; unit: Participants] | 48
Duration from diagnosis (Days) [Median (Inter-Quartile Range); unit: days] | 296 [76 to 855]

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Pain.
Description: Numerical Pain Rating Scale Total score 0-10 (0 is best outcome, 10 is worst outcome) 0-3 is mild pain, 4-7 is moderate pain, 7-10 is severe pain.
Time Frame: Approximately 12 wks from the baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale (0-10)
Arm/Group | Cancer Patients
Number analyzed (Participants) | 72
score on a scale (0-10) | 3 [1 to 5]

2. Secondary Outcome: Total Brief Pain Inventory (BPI)
Description: To assess the severity of pain and impact on functioning that included worst pain in last 24 hrs, least pain in last 24 hrs, pain average, pain right now, general activity, mood, walking ability, normal work, relationship with other, sleep and enjoyment of life.
  Each symptoms scales 0-10 (0 mean no symptom, not interfere, 10 mean most symptom, most interfere) total 70 scores
Time Frame: Approximately 12 wks from the baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cancer Patients
Number analyzed (Participants) | 72
score on a scale | 26 [8.5 to 40.5]

3. Secondary Outcome: Edmonton Symptom Assessment System(ESAS)
Description: To assess multi-directional of patients quality of life, included 9 symptoms ( pain,tired, neausea, depress, anxious, drowsiness, appetite, feeling of well being, shortness of breath) Each symptoms scales 0-9 (0 mean no Symptom, 9 mean most severe symptom) total ESAS 90 scores
Time Frame: Approximately 12 wks from the baseline
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Cancer Patients
Number analyzed (Participants) | 72
score on a scale | 23.5 [10.5 to 36.5]

4. Secondary Outcome: Percentage of Moderate to Severe Sedation
Description: Pasero Opioid-induced Sedation Scale (POSS)
  * S=sleep, easy to arouse
  * 1=awake/alert
  * 2= slight drowsy/easy aroused
  * 3=Frequently drowsy, arousable, drifts off to sleep during conversation
  * 4=Somnolent, minimal or no response to verbal and physical stimulation Score of 2-4 indicated moderate to severe sedation
Time Frame: Approximately 12 wks from the baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cancer Patients
Number analyzed (Participants) | 72
Participants | 6

5. Secondary Outcome: Percentage of Moderate to Severe Neausea and Vomitting
Description: Four points scale to evaluate opioid induce nausea and vomiting Total scales 0-3 (0 is best outcome, 3 is worst outcome)
  * 0= no nausea and vomiting
  * 1= mild symptom but not need any treatments. (only neausea)
  * 2= moderate symptom, need treatment, can control symptom. (have vomiting can control with medication)
  * 3= severe symptom, need treatment, cannot control symptom. (vomiting can not control with medication)
Time Frame: Approximately 12 wks from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cancer Patients
Number analyzed (Participants) | 72
Participants | 9

6. Secondary Outcome: Percentage of Moderate to Severe Constipation
Description: Stool free interval 72 (sfi72) to evaluate opioid induce costipation (OIC): 0-4.
  Total scale 0-4 (0 is best outcome, 4 is worst outcome)
  * 0 represented one defecation within the previous 72 hr
  * 1 denoted mild constipation (no defecation within the last 72 h)
  * 2 referred to the use of a maximum of 3 laxatives
  * 3 referred to the use of more than 3 laxatives
  * 4 referred to the use of all laxatives have failed Score of 2-4 indicated moderate to severe constipation
Time Frame: Approximately 12 wks from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Cancer Patients
Number analyzed (Participants) | 72
Participants | 17

7. Secondary Outcome: Percentage of Satisfied With the Service (Score=3)
Description: Satisfied score
  * 1=Dissatisfied
  * 2=Neutral
  * 3=Satisfied
Time Frame: Approximately 12 wks from the baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Cancer Patients
Number analyzed (Participants) | 72
Participants | 64

ADVERSE EVENTS:
Time Frame: We collected the adverse effect from pain medication such as sedation score, nausea and vomiting, constipation. from the baseline, FU1, FU2, FU3 (approximately 2-4 weeks eash interval) total 12 weeks.
Description: All cause mortality in this paper was 28 patients in 128 patients. The 28 patients died during the study duet to natural of disease. All patients were at risk because all of patients were diagnosed with cancer and 80% of patients were advanced stage of cancer. The 128 patients were number of patients who decided to treat in our clinic and our hospital during study time.
Arm/Group | Cancer Patients
All-Cause Mortality (participants affected / at risk) | 28/128
Serious Adverse Events (participants affected / at risk) | 0/128
Other Adverse Events (participants affected / at risk) | 32/128
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cancer Patients (N=128)
Moderate to severe sedation (Nervous system disorders) | 6
Moderate to severe nausea and vomiting (Gastrointestinal disorders) | 9
moderate to severe constipation (Gastrointestinal disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03474406/Prot_SAP_000.pdf